CLINICAL TRIAL: NCT06532292
Title: Physical Therapy Intervention for Pelvic Organ Prolapses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202401217DINC
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HIFEM (Experimental): During the initial appointment, participants will receive a comprehensive lifestyle advice leaflet covering pertinent information related to POP risk factors and guidance on diet, weight loss, the avoidance of heavy lifting, coughing, high-impact exercises. Following th educational component, participants will be asked to sit in an upright position at the center of an electromagnetic chair (such as the BTL EMSELLA, BTL Industries Inc., Boston MA) while remaining fully clothed for a duration of 28 minutes. To ensure optimal stimulation of the pelvic floor muscles, the physical therapist will carefully monitor the participant's chair posture throughout the treatment sessions and adjust the intensity of the electromagnetic stimulus according to the participant's tolerance threshold.
  Interventions: Device: HIFEM
- Biofeedback (Active Comparator): The biofeedback group will undergo PFMT with biofeedback and/or electrostimulation, administered twice a week over 8 weeks by a skilled physical therapist. During the biofeedback and electrical stimulation, participants will assume a supine position with a 45° angle of hip and knee flexion, refraining from actively contracting the PFMs. The intravaginal probe will be inserted into the vagina. The frequency of electrostimulation will be set between 10-50 Hz based on participant tolerance and the pulse duration will be adjusted to 300-500 μs. The stimulation intensity will be set at the maximum tolerable level. During biofeedback, participants will receive visual instructions to guide them in relaxing and contracting their PFMs.
  Interventions: Device: Biofeedback
- Usual care group (No Intervention): Participants allocated to the usual care (i.e., no physical therapy) group will receive the usual care provided by their obstetricians or gynecologists based on clinical judgment, in addition to the lifestyle advice leaflet provided by the research team. The lifestyle advice leaflet will be given to the participants immediately after the baseline assessment, and the usual care group will have no planned contact with the project staff until 8 weeks after the baseline assessment.

INTERVENTIONS:
Device: Biofeedback — To facilitate PFM function, electromyography biofeedback and electrical stimulation will be employed using an intravaginal probe, tailored to individual needs.
  Arms: Biofeedback
Device: HIFEM — The HIFEM device (i.e. BTL EMSELLA) is FDA approved and its indications are to provide entirely non-invasive electromagnetic stimulation of pelvic floor muscle for the purpose of rehabilitation of weak pelvic muscles and restoration of neuromuscular control for the treatment of male and female urinary incontinence.
  Arms: HIFEM

SUMMARY:
Pelvic floor muscle training (PFMT) and pessaries are first-line non-surgical conservative treatments for pelvic organ prolapse (POP). High-Intensity Focused Electromagnetic Field (HIFEM) is a noninvasive and painless device, designed to promote muscle strengthening and growth and has become a popular treatment option for urinary incontinence in the field of gynecology. However, HIFEM has not yet been rigorously compared to traditional physical therapy for POP. The objectives of this pilot study are to explore clinical effects of HIFEM on POP symptoms; to compare the effectiveness of HIFEM versus PFMT with biofeedback, and usual care on patient-centered outcomes; and to explore the acceptability of the interventions. This is a prospective, single-center randomized controlled trial with a nested qualitative interview study. Twenty-one women with POP, aged >20 years, will be recruited and randomly allocated to three groups, 'HIFEM' group, 'Biofeedback' group, and 'Usual care' group.The 'HIFEM' group will be asked to sit straight in the center of an electromagnetic chair and remained fully clothed for 28 minutes. The 'Biofeedback' group will receive PFMT with biofeedback and/or electrostimulation. Both 'HIFEM' and 'Biofeedback' groups will receive the interventions twice a week for 8 weeks. Participants allocated to the 'Usual care' group will receive the lifestyle advice leaflet only. All participants will be assessed for pelvic floor muscle function, symptom severity of POP, occurrence and distress related to pelvic floor dysfunction, and impact of pelvic floor dysfunction at baseline and immediately post-intervention.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is a prevalent, non-malignant condition affecting 30% to 50% women, with roughly 30% of these women undergo surgical intervention due to related symptoms impacting their daily lives. According to the international guidelines, the management of POP encompasses several approaches, including observation, lifestyle adjustments, pelvic floor muscle training (PFMT), the use of pessaries, reconstructive surgeries, obliterative surgeries, transperineal surgeries, and transabdominal surgeries. Among these, PFMT and pessaries are first-line non-surgical conservative treatments for POP. High-Intensity Focused Electromagnetic Field (HIFEM) is a noninvasive and painless device, designed to promote muscle strengthening and growth. Recently, the HIFEM has become a popular treatment option for urinary incontinence in the field of gynecology. The HIFEM, unlike traditional PFMT, does not require any exposure of the intimate part of the body; the patient is fully clothed and seated on the center of the chair during the treatment. However, while revolutionary, HIFEM has not yet been rigorously compared to traditional physical therapy for POP.

The objectives of this study are:

1. To explore clinical effects of HIFEM on POP symptoms.
2. To compare the effectiveness of HIFEM versus PFMT with biofeedback, and usual care on patient-centered outcomes.
3. To explore the acceptability of the interventions

This is a prospective, single-center randomized controlled trial with a nested qualitative interview study. Sixty-nine women with POP, aged >20 years, will be recruited and randomly allocated to three groups, 'HIFEM' group, 'Biofeedback' group, and 'Usual care' group. The 'HIFEM' group will be asked to sit straight in the center of an electromagnetic chair and remained fully clothed for 28 minutes. The process will be supervised by a female physical therapist who will also provide a lifestyle advice leaflet and education to the participants. The training will be provided at a frequency of two sessions per week over 8 weeks. The 'Biofeedback' group will receive PFMT with biofeedback and/or electrostimulation twice a week for 8 weeks with a physical therapist. Participants allocated to the 'Usual care' group will receive the lifestyle advice leaflet only. The baseline and immediately post-intervention assessments will include clinical examination of pelvic floor muscle function (digital palpation and transperineal ultrasound) and three questionnaires about symptom severity of POP, occurrence and distress related to pelvic floor dysfunction, and impact of pelvic floor dysfunction. This study will provide evidence of effectiveness of different modes of physical therapy program for women with POP and health-care professionals working with this population in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Women aged over 20 years
* Prolapse severity of stages 1, 2, or 3 in one or more compartments (anterior vaginal wall, uterine/cervical, vaginal vault, posterior vaginal wall)

Exclusion Criteria:

* Stage 4 prolapse
* Tumor in the pelvic region
* A recent surgical procedure (within 6 months)
* Metal implants
* Severe physical/psychiatric impairments
* Pregnancy or planning to become pregnant during the next 2 months
* Severe vaginal atrophy
* Vaginal infectious disease
* Neurologic disorders
* Receiving physical therapy treatments for prolapse or urinary incontinence
* Any contraindication listed in the investigational device manual

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2026-08-09 (Estimated)

PRIMARY OUTCOMES:
POP symptom severity | absolute values at baseline and 8 weeks
  The evaluation of POP symptom severity will utilize the Pelvic Organ Prolapse Symptom Score (POP-SS). The POP-SS comprises seven items gauging the frequency of various prolapse symptoms. Each item employs a five-point Likert scale response set (0-4). The cumulative scores of the seven questions result in a total score ranging from 0 to 28, where higher scores indicate more pronounced symptom severity.

SECONDARY OUTCOMES:
Distress related to pelvic floor dysfunction | absolute values at baseline and 8 weeks
  The distress related to pelvic floor dysfunction will be assessed using the Pelvic Floor Distress Inventory-20 (PFDI-20). This instrument consists of 20 questions in three domains: urinary (6 questions), POP (6 questions), and colorectal-anal (8 questions). The total score ranges from 0 - 300. Higher values indicate greater distress caused by pelvic floor dysfunction.
Impact of pelvic floor dysfunction | absolute values at baseline and 8 weeks
  The impact of pelvic floor dysfunction will be assessed using the Pelvic Floor Impact Questionnaire-7 (PFIQ-7). This questionnaire consists of seven questions in three domains (urinary, POP, and colorectal-anal). The total score ranges from 0 - 300. Higher scores indicate greater impact.
Pelvic floor muscle strength | absolute values at baseline and 8 weeks
  Digital measurement of squeeze and lift strength, recorded using the modified Oxford scale in lying and standing positions will be used. The Modified Oxford Scale quantifies pelvic floor muscle strength as 0, no contraction; 1, flicker; 2, weak; 3, moderate; 4, good; and 5, strong. Maximum voluntary contraction (MVC) strength will be measured over 3 seconds. Participants will need to repeat three MVC contractions, with a 3-second interval in between, and the best of three will be recorded.
Pelvic floor muscle endurance (time) | absolute values at baseline and 8 weeks
  Endurance will be measured by asking the participants to sustained an MVC for up to 10 seconds and the sustained time will be recorded in seconds.
Pelvic floor muscle endurance (repetition number) | absolute values at baseline and 8 weeks
  Endurance will also be measured by asking the participants to perform fast-twitch pelvic floor muscle contractions for up to 10 times with each MVC lasting 1 second. Endurance will be recorded as the number of time of fast contractions that the participant can execute.
Anteroposterior diameter of urogenital hiatus | absolute values at baseline and 8 weeks
  A real-time transperineal ultrasound, which will be used to measure the anteroposterior diameter of urogenital hiatus (mm) at rest, during PFM contraction (3 x 3-second contractions), and at maximum Valsalva (forced expiration against a closed glottis, with a relaxed pelvic floor, for at least 6 seconds).
Displacement of the bladder neck | absolute values at baseline and 8 weeks
  A real-time transperineal ultrasound, which will be used to measure the displacement of the bladder neck (mm) at rest, during PFM contraction (3 x 3-second contractions), and at maximum Valsalva (forced expiration against a closed glottis, with a relaxed pelvic floor, for at least 6 seconds).

OTHER OUTCOMES:
Acceptability of the intervention and the outcome measures | Immediately post-interventions
  Participants will be invited to participate in interviews about the acceptability of the intervention and the outcome measures. The semi-structured interview guide will guide the exploration of participants' experiences and perspectives on the interventions and outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Yin Lin, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The main reason for not sharing individual participant data is that the data are confidential.